CLINICAL TRIAL: NCT07237945
Title: Investigation of the Effects of Quadro-Iliac Plane Block and Wound Infiltration on Postoperative Acute Pain After Single-Level Lumbar Discectomy Surgery
Brief Title: Quadro-Iliac Plane Block Versus Wound Infiltration for Postoperative Pain After Single-Level Lumbar Discectomy
Status: Recruiting | Type: Observational
Sponsor: Elif Sarikaya Ozel (Other)
Responsible Party: Sponsor-Investigator, Elif Sarikaya Ozel, M.D., Karabuk University
Organization: Karabuk University (Other)
Other Study IDs: QIPB-LD2026
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain Management; Lumbar Discectomy; Regional Anaesthesia
Keywords: Quadro-Iliac Plane Block; Wound Infiltration; QIPB

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group QİPB: Patients receiving ultrasound-guided Quadro-Iliac Plane Block with 30 mL of 0.25% bupivacaine per side (total 60 mL) as part of routine postoperative analgesia after single-level lumbar discectomy.
- Group WI: Patients receiving ultrasound-guided wound infiltration with 20 mL of 0.25% bupivacaine into the surgical field at the end of surgery as part of routine postoperative analgesia after single-level lumbar discectomy.

SUMMARY:
This prospective observational study aims to compare the effects of the Quadro-Iliac Plane Block (QIPB) and wound infiltration (WI) on postoperative acute pain in adult patients undergoing elective single-level lumbar discectomy. QIPB is a newly introduced ultrasound-guided fascial plane block, and it is currently being used in routine clinical practice in our anesthesiology department as part of postoperative analgesia for lumbar spine surgery. Wound infiltration is a conventional method in which local anesthetic is injected into the surgical field at the end of the procedure.

In this study, eligible patients will be monitored prospectively without randomization or alteration of standard care. Postoperative pain scores, opioid consumption, nausea and vomiting, patient satisfaction, and recovery parameters will be evaluated during the first 24 hours after surgery. The study aims to provide real-world clinical evidence comparing these two analgesic techniques in lumbar discectomy patients.

DETAILED DESCRIPTION:
This prospective observational study aims to evaluate and compare the postoperative analgesic outcomes of two routinely used analgesic techniques-Quadro-Iliac Plane Block (QIPB) and wound infiltration (WI)-in adult patients undergoing elective single-level lumbar discectomy. Both QIPB and WI are standard components of postoperative pain management in our hospital, and the type of analgesic technique administered to each patient is determined solely by the attending anesthesiologist based on routine clinical judgment. The research team does not influence clinical decision-making, perform block procedures, or modify any aspect of patient care. All interventions included in this study reflect standard institutional practice.

The primary objective is to compare cumulative opioid consumption during the first 24 hours after surgery between patients receiving QIPB and those receiving WI. Secondary objectives include evaluating postoperative pain scores, early recovery parameters, patient satisfaction, postoperative nausea and vomiting (PONV), rescue analgesic requirements, block-related complications, and hospital length of stay.

Clinical Routine and Analgesic Protocol

All patients will be managed according to the standard multimodal analgesia protocol routinely used in our neurosurgery operating room. Intraoperatively, intravenous tenoxicam 20 mg, tramadol 100 mg and dexamethasone 8 mg will be administered as part of routine analgesic and antiemetic care. Paracetamol 1 g IV will be given at the end of surgery and continued at regular intervals postoperatively. Rescue analgesia will consist of intravenous tramadol 100 mg infused over 30 minutes, with a maximum daily dose of 300 mg; if pain remains uncontrolled (NRS ≥4). All patients will receive intravenous morphine patient-controlled analgesia (Body Guard 575 Pain Manager) with a standard setting of 1 mg bolus dose, a 10-minute lockout interval, and a 4-hour limit set to 80% of the maximum allowable dose.

Block Techniques (Performed as Part of Routine Care)

QIPB Group:

QIPB is a newly introduced interfascial block technique currently used in our clinic for postoperative lumbar spine analgesia. At the end of surgery and before extubation, the patient is placed in the prone position. A low-frequency convex ultrasound probe (2-6 MHz) is positioned at the L3 midline in the transverse plane to identify the spinous process. The probe is then moved laterally and caudally to visualize the attachment of the quadratus lumborum muscle to the iliac crest. Under ultrasound guidance, a 22G, 100-mm block needle is advanced into the fascial plane between the quadratus lumborum and erector spinae muscles. A total of 60 mL of 0.25% bupivacaine (30 mL per side) is injected bilaterally. The procedure is performed by experienced anesthesiologists as part of normal clinical practice.

Wound Infiltration Group (WI):

WI is a routine analgesic method performed in our operating room. At the end of surgery, before skin closure, 20 mL of 0.25% bupivacaine is infiltrated into the surgical field in multiple tissue layers. This procedure is performed entirely according to the attending anesthesiologist's habitual clinical practice.

Postoperative Assessment

Postoperative pain will be assessed using the 11-point Numeric Rating Scale (NRS; 0-10) at rest and during movement (deep breathing or coughing) at 0, 3, 6, 12, and 24 hours after surgery. PONV will be evaluated using a verbal descriptive scale. If PONV score is ≥3, 4 mg IV ondansetron will be administered. Patient satisfaction and quality of recovery will be assessed using the Turkish version of the QoR-15 questionnaire preoperatively, on postoperative day 1, and at discharge.

Block-related complications (hematoma, bleeding at the injection site, LAST), opioid-related side effects (itching, sedation, respiratory depression), time to first PCA demand, time to first mobilization, rescue analgesic requirements, and hospital length of stay will be recorded.

All data will be analyzed using SPSS software. Statistical tests will be selected based on data distribution, and a p-value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 80 years
* Scheduled for elective single-level lumbar discectomy
* ASA physical status I-III
* Able to use patient-controlled analgesia (PCA)
* Able and willing to provide written informed consent

Exclusion Criteria:

* History of opioid use for longer than 4 weeks
* Presence of chronic pain before surgery (e.g., migraine, fibromyalgia)
* Alcohol or substance dependence
* Known allergy or hypersensitivity to local anesthetics or opioids
* Significant organ dysfunction (e.g., severe hepatic or renal disease)
* Revision or multilevel spine surgery
* Contraindications to regional anesthesia
* Severe psychiatric disorders limiting cooperation (e.g., psychosis, dementia)
* Pregnancy or breastfeeding
* Hematologic disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled to undergo elective single-level lumbar discectomy at Karabuk Training and Research Hospital. Eligible participants will be evaluated preoperatively and enrolled prospectively according to predefined inclusion and exclusion criteria. No healthy volunteers are included.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
24-hour cumulative opioid consumption | postoperative day 1
  Total opioid consumption within the first 24 hours, including PCA-administered morphine and rescue analgesics converted to morphine milligram equivalents (MME).

SECONDARY OUTCOMES:
12-hour cumulative opioid consumption | postoperative 12th hour
  Total opioid consumption within the first 12 hours, including PCA-administered morphine and rescue analgesics converted to MME.
Block performance time | intraoperative period
  Total time (minutes) required to complete the QIPB procedure.
Postoperative pain scores (NRS at rest and activity) | postoperative day 1
  Pain status at rest and while activity will be assessed by numeric rating scale (NRS) score at 0, 3, 6, 12, 18 and 24 hours after surgery. In addition, the time until the first analgesic requirement will be recorded. The NRS is an 11-point numeric scale that ranges from 0 to 10.
Patient-reported quality of recovery (QoR-15 score) | Postoperative day 1 and at postoperative day 2-4 day
  Quality of recovery assessed using the validated 15-item QoR-15 questionnaire.
Postoperative nausea and vomiting incidence (PONV) | Postoperative day 1
  The severity of postoperative nausea and vomiting (PONV) will be assessed using a descriptive verbal rating scale at 0, 3, 6, 12, 18 and 24 hours after extubation. If a score of 3 or more, ondansetron 4 mg IV will be administered and will repeat after 8 hours if required (The PONV scale is 0 = no nausea; 1 = slight nausea; 2 = moderate nausea; 3 = vomiting once; and 4 = vomiting more than once).
Time to first PCA analgesic demand | Postoperative day 1
  Time at which the first analgesic is requested
Number of patients requiring rescue analgesia | Postoperative day 1
  Number of patients who required rescue analgesia despite PCA use.
Time to first mobilization | Postoperative day 2-4
  Time (hours) from the end of surgery to first assisted ambulation with a physiotherapist.
Block-related complications | Postoperative day 7
  Incidence of complications such as bleeding, hematoma, or local anesthetic systemic toxicity (LAST).
Opioid-related adverse effects | Postoperative day 7
  Presence of itching, sedation, fatigue, or respiratory depression related to opioid use.
Length of hospital stay | Postoperative day 2-4
  Duration of hospitalization measured in hours or days.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Sarikaya Ozel, Principal Investigator — Karabuk Training and Research Hospital, Department of Anesthesiology
Locations (1):
- Karabuk Training and Research Hospital, Department of Anesthesiology and Reanimation, Karabük, Turkey (Türkiye)